CLINICAL TRIAL: NCT06777667
Title: Impact of Resilience and Family Dynamics on Disease Severity in Women With Fibromyalgia: Comparison With Healthy Controls
Brief Title: Fibromyalgia Severity: Role of Resilience and Family Dynamics
Acronym: FSRRFD
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AntalyaCityHospital
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Fibromyalgia; Resilience
Keywords: Fibromyalgia; Connor-Davidson Resilience Scale
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fibromyalgia group: Individuals diagnosed with fibromyalgia according to the 2016 ACR criteria. Participants will be recruited from the Physical Medicine and Rehabilitation Clinic at Antalya City Hospital.
  Inclusion Criteria:
  Female, aged 25-45 years Diagnosis of fibromyalgia according to the 2016 revision of 2010/2011 ACR criteria Able to provide informed consent
- Healthy control group: Age- and sex-matched healthy female individuals. No diagnosis of fibromyalgia or any other chronic pain condition. Recruited from the community or other appropriate sources.
  Inclusion Criteria:
  * Female, aged 25-45 years
  * No history of fibromyalgia or other chronic pain conditions
  * Able to provide informed consent

SUMMARY:
This cross-sectional survey study aims to examine the resilience and family dynamics between newly diagnosed fibromyalgia (FM) patients and healthy individuals. The study will analyze demographic data including parental attitude and childhood trauma and resilience levels using the Connor-Davidson Resilience Scale (CD-RISC-10) in fibromyalgia patients and healthy controls. The Revised Fibromyalgia Impact Questionnaire (FIQR) will also be administered to FM patients to determine the total impact and severity of the disease (mild, moderate, severe, very severe). In addition to aiming to reveal how FM patients compare to healthy individuals in terms of resilience and parental attitude, this study will also examine the relationship between disease severity and these psychosocial variables. As a result, the data obtained are expected to reveal both potential differences in resilience and family problems in FM patients and the relationship of these factors with disease severity.

DETAILED DESCRIPTION:
FM is a common disease worldwide, characterized by chronic widespread pain, sleep problems, physical fatigue, and cognitive difficulties. It is estimated that symptoms are seen in around 2-4% of the population. Although FM is due to a complex disease model triggered by biological and psychosocial variables, the details are still unclear.

While psychological resilience plays a critical role in coping with stress and chronic pain, a supportive family environment can contribute to individuals developing effective coping mechanisms. Research shows that low resilience levels can trigger FM and a controlling family environment can negatively affect emotional functioning.

The increase in the incidence of FM in recent years has placed additional burdens on the healthcare system. Therefore, it is necessary to provide new perspectives that will guide clinicians who face FM and contribute to improving treatment processes.

The research aims to develop a deep understanding of the etiology and course of FM, as well as to contribute to customizing individual treatment approaches and health services by revealing the effects of psychosocial factors. This study will contribute to the understanding of the relationships between psychological resilience, family dynamics and disease severity in fibromyalgia patients. The data to be obtained will help develop new perspectives and suggestions for clinical practices by emphasizing the importance of psychological support and family dynamics in the treatment processes of fibromyalgia. In addition, comparisons with healthy controls may lead to a better understanding of the needs of individuals with FM. Another important benefit expected from the study is to place more emphasis on the importance of resilience and problems in child development. These studies have the potential to reduce the risks of developing FM and similar diseases in tomorrow's adults. In this context, primary prevention strategies may contribute to public health and the burden on the health system.

This study aims to examine the relationships between psychological resilience, childhood problems and severity of fibromyalgia symptoms between FM patients and healthy control groups. In particular, it was aimed to determine which elements significantly affect symptom severity by evaluating the effects of these factors on FM.

The hypotheses of the study:

Hypothesis 1: Individuals with low psychological resilience and a negative parental attitude during childhood will experience more severe FM symptoms.

Hypothesis 2: FM patients will have lower psychological resilience and more negative parental attitude compared to healthy controls.

Rationale for the study:

FM is a common disease characterized by chronic widespread pain, sleep problems, physical fatigue, and cognitive difficulties. It is characterized by chronic widespread pain, somatic symptoms, and cognitive difficulties. FM is seen in all populations worldwide, and the prevalence of symptoms varies between 2% and 4% in the general population. A model has been proposed for the pathogenesis of FM in which biological and psychosocial variables influence the susceptibility, triggering, and worsening of a chronic disease, but the details are unclear.

FM is a complex and multifactorial disorder, and the severity of its symptoms may be affected by the individual's psychosocial circumstances. While psychological resilience plays a critical role in coping with chronic pain and stress, a supportive family environment may encourage individuals to develop effective coping mechanisms. There may be a link between FM and resilience, as resilience is closely related to an individual's response to acute or chronic stress, which can affect chronic pain conditions such as FM. Resilience is a complex structure that is contributed by genetics and environmental factors, and in some individuals, these factors may help to develop a personality that is more resilient to stressful life events. Therefore, low resilience may be a trigger for FM. The family environment may also be a factor contributing to the complex structure of fibromyalgia. Previous research has found that a controlling (highly regimented and less independent) family environment in early adolescence is a key factor predicting poorer long-term emotional functioning in juvenile FM patients. Reports indicate that the incidence of fibromyalgia increased from 2001 to 2013, suggesting that the healthcare system will be further burdened by the management of this disease. This study will provide important guidance for clinicians facing FM and will help to provide new perspectives on the management of the disease.

This study aims to better understand the potential contributions and effects of these factors on the health of individuals by examining the effects of psychological resilience and family environment on the severity of fibromyalgia. The findings to be obtained in these areas may contribute to the development of individual treatment approaches and the customization of health services.

This study will provide data that can help improve treatment processes by developing a deeper understanding of the etiology and course of FM. In addition, understanding the role of psychosocial and environmental factors will allow the development of more targeted interventions for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: Women between the ages of 25-45.
2. Diagnosis: For fibromyalgia Group: Individuals diagnosed according to the 2016 revision of the American College of Rheumatology's 2010/2011 fibromyalgia diagnostic criteria. For healthy Control Group: Healthy women without a fibromyalgia diagnosis.
3. Consent: Individuals who volunteered to participate in the research processes and gave informed consent regarding the details of participation and signed the consent form.

Exclusion Criteria:

1. Serious medical conditions: Individuals with serious health problems such as autoimmune diseases, cancer, severe heart and lung diseases, or acute pain caused by trauma, surgery, inflammatory joint diseases, etc.
2. Psychiatric conditions: Individuals with psychiatric diseases, medication use, or whose mental state may affect their ability to understand and complete the survey questions.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — "Female" refers to individuals who identify as female.
Study Population: The study population will include adult females aged 25-45 years. Participants will be divided into two groups: (1) individuals with a diagnosis of fibromyalgia and (2) healthy female controls within the same age range. All participants will be recruited through convenience sampling, such as patients visiting the Physical Medicine and Rehabilitation Clinic at Antalya City Hospital, and will provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Resilience levels | Baseline/ at the time of enrollment
  Comparison of resilience scores between fibromyalgia patients and healthy controls. (Resilience was measured using the 10-item Connor Davidson- Resilience Scale, which ranges from 0 to 40, with higher scores reflecting greater resilience and better psychological adaptability.)

SECONDARY OUTCOMES:
Correlation between resilience and the severity of fibromyalgia symptoms. | Baseline/ at the time of enrollment
  Resilience scores in relation to the severity of fibromyalgia symptoms. (Severity of fibromyalgia symptoms was assessed using the Revised fibromyalgia Impact Questionnaire, which measures functional impairment, overall impact, and symptom severity in fibromyalgia patients. The total score ranges from 0 to 100, with higher scores reflecting greater disease burden and worse functional status.)

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Duman Sahin, MD, Study Chair — Physical Medicine and Rehabilitation
Locations (1):
- Antalya City Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hauser W, Ablin J, Fitzcharles MA, Littlejohn G, Luciano JV, Usui C, Walitt B. Fibromyalgia. Nat Rev Dis Primers. 2015 Aug 13;1:15022. doi: 10.1038/nrdp.2015.22. PMID 27189527
- [Background] Casale R, Sarzi-Puttini P, Botto R, Alciati A, Batticciotto A, Marotto D, Torta R. Fibromyalgia and the concept of resilience. Clin Exp Rheumatol. 2019 Jan-Feb;37 Suppl 116(1):105-113. Epub 2019 Feb 8. PMID 30747098
- [Background] Sil S, Lynch-Jordan A, Ting TV, Peugh J, Noll J, Kashikar-Zuck S. Influence of family environment on long-term psychosocial functioning of adolescents with juvenile fibromyalgia. Arthritis Care Res (Hoboken). 2013 Jun;65(6):903-9. doi: 10.1002/acr.21921. PMID 23281206
- [Background] Collin SM, Bakken IJ, Nazareth I, Crawley E, White PD. Trends in the incidence of chronic fatigue syndrome and fibromyalgia in the UK, 2001-2013: a Clinical Practice Research Datalink study. J R Soc Med. 2017 Jun;110(6):231-244. doi: 10.1177/0141076817702530. Epub 2017 Mar 30. PMID 28358988
- [Background] Bennett RM, Friend R, Jones KD, Ward R, Han BK, Ross RL. The Revised Fibromyalgia Impact Questionnaire (FIQR): validation and psychometric properties. Arthritis Res Ther. 2009;11(4):R120. doi: 10.1186/ar2783. Epub 2009 Aug 10. PMID 19664287
- [Background] Ediz L, Hiz O, Toprak M, Tekeoglu I, Ercan S. The validity and reliability of the Turkish version of the Revised Fibromyalgia Impact Questionnaire. Clin Rheumatol. 2011 Mar;30(3):339-46. doi: 10.1007/s10067-010-1546-8. Epub 2010 Aug 12. PMID 20703890
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Background] Fowler PC. Factor structure of the Family Environment Scale: effects of social desirability. J Clin Psychol. 1982 Apr;38(2):285-92. doi: 10.1002/1097-4679(198204)38:23.0.co;2-9. PMID 7068862